CLINICAL TRIAL: NCT05341583
Title: A Phase Ⅲ, Double-blind, Randomized, Placebo-Controlled Study to Assess the Efficacy and Safety of Ensartinib Versus Placebo as Adjuvant Therapy in Patients With Anaplastic Lymphoma Kinase (ALK)-Positive Stage IB- IIIB Non-small Cell Lung Cancer.
Brief Title: Ensartinib as Adjuvant Treatment in Anaplastic Lymphoma Kinase (ALK) Positive Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTP-42338
Record Dates: First submitted 2022-04-18; First posted 2022-04-22 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ensartinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ensatinib (Experimental): Ensatinib ( 225 mg, once daily), in accordance with the randomization schedule
  Interventions: Drug: Ensartinib
- Placebo (Placebo Comparator): Placebo ( 225 mg, once daily), in accordance with the randomization schedule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ensartinib — Ensartinib 225 mg once daily until disease recurrence or up to 2 years, whichever occurs earlier.
  Other Names: X-396
  Arms: Ensatinib
Drug: Placebo — Placebo 225 mg once daily until disease recurrence or up to 2 years, whichever occurs earlier.
  Arms: Placebo

SUMMARY:
This double-blind, randomized, placebo-controlled, multicenter, Phase III study is designed to evaluate the efficacy and safety of ensatinib compared with placebo as adjuvant treatment in ALK positive stage II-IIIB non-small cell lung cancer after surgical resection with or without chemotherapy.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled, multicenter, Phase III study, the primary endpoint is disease-free survival. Participants in the experimental arm will receive Ensatinib at 225 mg orally once a day taken with or without food for 2 years. Participants in the control arm will receive placebo at 225 mg orally once a day taken with or without food for 2 years. Treatments will continue until disease recurrence, meeting one of treatment discontinuation criteria (eg, patient decision, adverse event, pregnancy), or achieving a maximum treatment duration of 2 years, whichever occurs earlier. At the time of treatment discontinuation, participants will enter a survival follow-up until death, withdrawal of consent or study closure, whichever occurs earlier.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of primary non-small cell carcinoma of the lung.
* Patients must be classified post-operatively as Stage IB-IIIB(T3N2M0) on the basis of pathologic criteria after complete surgical resection(R0).
* Complete recovery from surgery and standard post-operative therapy (if applicable) at the time of randomization.
* Confirmation by the central laboratory that the tumour harbours ALK positive.
* At least 1-year life expectancy.
* Eastern Cooperative Group (ECOG) Performance Status score of 0 or 1.
* The laboratory test values should meet the following requirements:

  1. Absolute neutrophil count ≥ 1.5 x 109/L , Platelets ≥ 100 x 109/L ，hemoglobin ≥9g/dL
  2. Total bilirubin≤ 1.5 x institutional upper limit of normal,AST and ALT≤ 2.5 x institutional upper limit of normal
  3. Creatinine≤ 1.5 x institutional upper limit of normal ,if not, Creatinine Clearance ≥ 50 ml/min
  4. International normalized ratio (INR) and prothrombin time ≤1.5 x institutional upper limit of normal; and activated partial thromboplastin time (aPTT) ≤1.5 x institutional upper limit of normal
* Female patients must have a negative pregnancy test at baseline.

Exclusion Criteria:

* Patients who are participating in other clinical studies or are receiving other investigational drugs , or investigational devices within 4 weeks before the first dose of our study drugs. If patients are participating in non-interventional clinical trials, they can be included in this study.
* Patients who have a presence of unresectable or metastatic disease, the pathological diagnosis show the microscopically positive surgical margins or extranodal invasion, or residual disease of surgery，or had only segmentectomies or wedge resections.
* Patients with superior sulcus cancer.
* Patients who have received a surgery with total right lung resection.
* History of other malignancies within 5 years of the first dose of the study drug, except: malignant tumors that can be expected to recover after treatment.
* Prior treatment with other anti-cancer treatments or NSCLC including chemotherapy, radiotherapy, targeted therapy (such as small molecule tyrosine kinase inhibitors targeting EGFR, VEGFR or other pathways, monoclonal antibodies, etc.), immunotherapy, investigational therapy, etc. but except platinum based chemotherapy for adjuvant therapy.
* Major surgery within 3 weeks of the first dose of the study drug.
* Patients who have used traditional Chinese medicines and traditional Chinese medicine preparations with indications for anti-tumor therapy or adjuvant therapy for tumors within 14 days of the first dose of the study drug.
* Patients who have used the following drugs within 14 days before the first dose : strong inhibitors, strong inducers of CYP3A or CYP3A substrates with a narrow therapeutic index.
* Patients who have severe cardiovascular disease.
* Patients with a known allergy to Tartrazine，a dye used in 100mg capsules.
* Severe active infection, interstitial lung disease/pneumonitis, or any serious underlying disease that may interfere with the subject's treatment with the regimen within 2 weeks prior to the first dose of study drug.
* Active HIV virus antibody,Treponema pallidum antibody positive.
* Active hepatitis B, hepatitis C virus antibody positive, or active tuberculosis.
* Presence of active gastrointestinal (GI) disease or other conditions that will interfere significantly with the absorption, distribution, metabolism, or excretion of study drugs.
* According to the judgment of the investigator, other conditions may affect the compliance of the protocol or affect the subject's signing of the informed consent, or is not suitable for participating in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-23 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) | up to 5 years
  From date of randomization until date of tumor recurrence or death, whichever occurs earlier

SECONDARY OUTCOMES:
DFS rate at 3 years | Assessed at 3 years
DFS rate at 5 years | Assessed at 5 years
Overall survival (OS) | Assessed at 5 years
OS rate at 5 years | up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- TianJin Medical University Cancer Institute & Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No